CLINICAL TRIAL: NCT02183324
Title: A Randomised, Double-blind, Placebo-controlled, Multiple Dose Phase II Study of BI 1356 BS (0.5 mg, 2.5 mg, and 10 mg in Tablet q.d. Administered Orally for 28 Days) to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: BI 1356 BS in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.12
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (4):
- Low dose of BI 1356 BS (Experimental)
  Interventions: Drug: Low dose of BI 1356 BS
- Medium dose of BI 1356 BS (Experimental)
  Interventions: Drug: Medium dose of BI 1356 BS
- High dose of BI 1356 BS (Experimental)
  Interventions: Drug: High dose of BI 1356 BS
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of BI 1356 BS
  Arms: Low dose of BI 1356 BS
Drug: Medium dose of BI 1356 BS
  Arms: Medium dose of BI 1356 BS
Drug: High dose of BI 1356 BS
  Arms: High dose of BI 1356 BS
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BI 1356 BS (0.5 mg, 2.5 mg, and 10 mg) administered orally once daily for 28 days in Japanese patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with a diagnosis of type 2 diabetes mellitus treated with diet and/or exercise only or with one or two oral hypoglycaemic agents except glitazones
* Glycosylated haemoglobin A1 (HbA1c)

  * <= 8.5% at screening for patients treated with diet and/or exercise and/or one oral hypoglycaemic agent or
  * <= 8.0% at screening for patients treated with two oral hypoglycaemic agents
* Age ≥21 and ≤ 70 years
* BMI ≥ 17.6 and ≤ 35 kg/m2

Exclusion Criteria:

* Any finding of the medical examination including blood pressure, pulse rate and electrocardiogram (ECG) deviating from normal and of not acceptable clinical relevance
* Clinically relevant concomitant diseases like renal insufficiency, cardiac insufficiency (NYHA II-IV), known cardiovascular diseases including hypertension (>150/95 mmHg), stroke, and transient ischemic attack (TIA).
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, except for type 2 diabetes mellitus, hyperlipidaemia and medically treated hypertension
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or relevant neurological disorders except polyneuropathy
* Chronic or relevant acute infections (e.g., human immunodeficiency virus (HIV), hepatitis)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug before drug administration except anti-hypertensives, acetylsalicylic acid, and statins
* Use of drugs decreasing blood glucose within 10 days before drug administration
* Participation in another trial with an investigational drug within two months before drug administration
* Alcohol abuse
* Drug abuse
* Blood donation (100 mL or more within four weeks before drug administration)
* Excessive physical activities (within one week before drug administration or during the trial)
* Any laboratory value outside the reference range and the clinical relevance is not acceptable (or the value is more than three times higher than the upper limit of the normal range, e.g., liver enzymes such as aspartate aminotransferase (AST(serum glutamate oxaloacetate transaminase/ SGOT)), alanine transaminase (ALT(serum glutamate pyruvate transaminase/ SGPT)), alkaline phosphatase (γALP), and lactate dehydrogenase (LDH)
* Fasted blood glucose >240 mg/dL (=13.3 mmol/L) on two consecutive days during washout
* Serum creatinine above 1.3 mg/dL at screening
* Pregnancy or child-bearing potential patients and breast-feeding patients
* Not willing to use adequate contraception (condom use plus another form of contraception, e.g., spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until one month after the last intake

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-02; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Global assessment of tolerability by the investigator on a 4-point scale (good, satisfactory, not satisfactory and bad) | Day 43
Number of patients with adverse events | Up to day 50
Number of patients with clinically relevant changes in vital signs (blood pressure, pulse rate) | Up to day 50
Number of patients with clinically relevant changes in clinical laboratory tests (haematology, clinical chemistry, and urinalysis) | Up to day 50

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) at different time points | Up to day 43
Time from last dosing to the maximum concentration of the analyte in plasma (tmax) at different time points | Up to day 43
Area under the concentration time curve of the analyte in plasma (AUC) at different time points | Up to day 43
Amount of the analyte that is eliminated in urine (Ae) at different time points | Up to day 43
Fraction of parent drug eliminated in urine (fe) at different time points | Up to day 43
Renal clearance of the analyte (CLR) at different time points | Up to day 43
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | After the last dose on day 28 up to day 43
Average concentration of the analyte in plasma at steady state (Cavg) | After the last dose on day 28 up to day 43
Terminal half-life of the analyte in plasma at steady state (t1/2,ss) | After the last dose on day 28 up to day 43
Terminal rate constant in plasma at steady state (λz,ss) | After last dose on day 28 up to day 43
Mean residence time of the analyte in the body at steady state after oral administration (MRTpo,ss) | After last dose on day 28 up to day 43
Apparent clearance of the analyte in plasma at steady state after extravascular multiple dose administration (CL/F,ss) | After last dose on day 28 up to day 43
Apparent volume of distribution during the terminal phase λz at steady state following extravascular administration (Vz/F,ss) | After last dose on day 28 up to day 43
Predose concentration of the analyte in plasma (Cpre) at different time points immediately before administration of the Nth dose | Up to day 28
Calculation of accumulation ratio of the analyte in plasma based on Cmax (RA,Cmax) | Up to day 43
Calculation of accumulation ratio of the analyte in plasma based on AUCτ (RA,AUCτ) | Up to day 43
Minimum dipeptidyl peptidase IV (DPP-IV) activity (Emin) at different time points | Up to day 43
Time to reach minimum DPP-IV activity (tmin) at different time points | Up to day 43
DPP-IV activity at different time points | Up to day 43

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24393553